CLINICAL TRIAL: NCT06298500
Title: Retrospective, Single Center Clinical Study on the Clinical Performance of Histoacryl® Lapfix - Cannula for Laparoscopic Inguinal Hernia Repair
Brief Title: Clinical Performance of HISTOACRYL® LAPFIX - CANNULA for Laparoscopic Inguinal Hernia Repair
Acronym: HISTOLAP
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2115
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Inguinal Hernia
Keywords: laparoscopic mesh fixation; inguinal hernia repair surgery; Cyanoacrylate; Histoacryl®
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Histoacryl Lapfix: Histoacryl Lapfix - Cannula for laparoscopic mesh fixation in patients undergoing hernia repair surgery
  Interventions: Device: hernia repair surgery

INTERVENTIONS:
Device: hernia repair surgery — In recent years, atraumatic mesh fixation with tissue adhesive has increasingly become the method of choice. It is the recommended mesh fixation method by the International Hernia Society Guidelines. In this study patients with inguinal hernia are treated by placing a prosthetic mesh in one of the layers of the abdominal wall to cover the weakness, the mesh is fixed by Histoacryl LapFix,
  Other Names: laparoscopic mesh fixation with Histoacryl Lapfix - Cannula

SUMMARY:
The goal of this retrospective study is to identify the incidence of hernia recurrence following the application of Histoacryl® Lapfix - Cannula for laparoscopic mesh fixation in patients undergoing hernia repair surgery. All adult patients who underwent laparoscopic inguinal hernia repair with Histoacryl® Lapfix - Cannula in the period June 2018 - March 2021 at Hospital San Juan de Dios will be analysed. The investigator team will access electronical medical records for the cohort of patients identified.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* treated between June 2018 and March 2021 at the Hospital San Juan de Dios for laparoscopic mesh fixation with Histoacryl Lapfix - Cannula after inguinal hernia repair surgery.

Exclusion Criteria:

* No exclusion criteria has been set.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) treated in the period June 2018 to March 2021 at the Hospital San Juan de Dios for laparoscopic mesh fixation with Histoacryl Lapfix - Cannula after inguinal hernia repair surgery.
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence rate | until 6 months postoperatively
  Describe the incidence of hernia recurrence following the application of Histoacryl® LapFix - Cannula for laparoscopic mesh fixation in patients undergoing hernia repair surgery. The incidence of hernia recurrence is documented from the medical records until 6 months postoperatively.

SECONDARY OUTCOMES:
Delayed tissue adhesive polymerization | intraoperatively
  The polymerization time of Histoacryl® (about 30 seconds) takes longer than expected.
Intraoperative bleeding requiring therapeutic measures | intraoperatively
  Bleeding that requires additional measures than normal practice for stopping the hemorrhage.
Organ injury | intraoperatively
  Cumulative Number of patients suffering from Injury of an organ adjacent to the defect.
Hernia recurrence | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of Hernia recurring again after repair
Mesh migration | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients in whom Mesh has moved from its original position
Adhesions | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients in whom tissue is adhered and allows no physiological movement
Erosion | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from a mesh erosion into the bladder/urethra include painful voiding, urinary frequency, urgency, hematuria, recurrent urinary tract infection, urinary calculi and urinary fistula.
Meshoma formation | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from a wrinkling of the mesh that causes pain or hernia recurrence. Nerve entrapment or damage. Rejection of the mesh implant.
Tack hernias | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients requiring tack fixation was needed
Surgical Site Infection (superficial, deep, intraabdominal) | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from Surgical Site Infection classified according on Center for Disease Control and Prevention criteria (A1: superficial, A2: deep, A3:
  organ/space)
Hematoma | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from a solid swelling of clotted blood within the tissues.
Seroma | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from a mass or lump caused by a buildup of clear fluid in a tissue, organ or body cavity
Hemorrhage | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from an escape of blood from a ruptured blood vessel.
Orchitis | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of patients suffering from inflammation of the testicles
Other Adverse Event | at discharge and 1 month postoperatively. There is the possibility to extend the follow-up period until 6 months
  Cumulative Number of any other adverse event not mentioned.
Reintervention | until 6 months postoperatively
  Patient requiring to be operated again for any reason.
Mesh repositioning or removal | until 6 months postoperatively
  Patient requiring being operated again for repositioning or removal of the Mesh
Acute or chronic pain | until 6 months postoperatively
  pain persisting beyond 6 months postoperatively re-quiring analgesic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Juan de Dios, Santa Cruz de Tenerife, Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No